CLINICAL TRIAL: NCT03983681
Title: Evaluation of a Theory-Driven Manualized Approach to Improving New Learning and Memory in MS
Acronym: STEM
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Kessler Foundation (Other)
Responsible Party: Principal Investigator, Nancy Chiaravalloti, Director, Kessler Foundation
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: R-1045-18
Record Dates: First submitted 2019-06-10; First posted 2019-06-12 (Actual); Last update posted 2025-05-07 (Actual); Status verified 2025-05

CONDITIONS: Multiple Sclerosis
Keywords: Multiple Sclerosis; MS; Relapsing-Remitting MS; Progressive MS; RRMS; PPMS; SPMS; Primary Progressive; Secondary Progressive
MeSH Terms: conditions — Multiple Sclerosis

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Masking Description: Participants will be blind as to which treatment group they are being placed. Study staff conducting baseline and follow-up assessments will also be blind as to which group participants are placed. Study staff conducting intervention sessions will be blind to participants' baseline and follow-up assessment performance.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Experimental (Experimental): The experimental group will receive memory enhancement exercises administered twice a week for 4 weeks (8 training sessions).
  Interventions: Behavioral: Strategy-Based Training to Enhance Memory (STEM)
- Control group (Placebo Comparator): The control group will receive placebo memory enhancement exercises administered twice a week for 4 weeks (8 training sessions).
  Interventions: Behavioral: Placebo control exercises

INTERVENTIONS:
Behavioral: Strategy-Based Training to Enhance Memory (STEM) — Protocol designed to improve memory functioning in individuals with neurological injuries administered for 4 weeks (8 training sessions).
  Arms: Experimental
Behavioral: Placebo control exercises — Placebo control memory exercises will be administered for 4 weeks (8 training sessions).
  Arms: Control group

SUMMARY:
The purpose of this research study is to investigate the effectiveness of a memory enhancement technique in persons with Multiple Sclerosis.

DETAILED DESCRIPTION:
The purpose of this research study is to investigate the effectiveness of a memory enhancement technique in persons with Multiple Sclerosis (MS). The study is designed to research how well this technique can help people with MS improve their memory and their ability to function better in everyday life.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of Multiple Sclerosis
* Ability to read and speak English fluently
* Difficulties with learning and memory skills

Exclusion Criteria:

* Prior diagnosis of stroke or other neurological injury/disease
* Flare up of symptoms within a month of study participation
* History of significant psychiatric illness (e.g., bipolar disorder, schizophrenia, psychosis) or current diagnosis of Major Depressive Disorder, Schizophrenia, Bipolar Disorder I or II
* Current significant alcohol or substance abuse
* Taking exclusionary medication (study team will review medications)

For Optional MRI:

* Pacemaker or other implanted electrical device, brain stimulator, aneurysm clip (metal clips on the wall of a large artery), metallic prostheses (including metal pins and rods, heart valves, and internal hearing aids [cochlear implants]), permanent eyeliner, implanted delivery pumps, or shrapnel fragments.
* Dental implants
* Left-handed

Ages: 18 Years to 59 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 120 (Estimated)
Dates: Start 2019-09-26 (Actual); Primary Completion 2025-09-15 (Estimated); Study Completion 2025-09-30 (Estimated)

PRIMARY OUTCOMES:
Changes in scores on self-report measure of everyday cognition (subjective) | Baseline (week 1), immediately post-intervention (week 6) and long-term follow-up (week 6 months post-intervention)
  Perceived Deficits Questionnaire
Changes in scores on self-report measure of everyday cognition (objective) | Baseline (week 1), immediately post-intervention (week 6) and long-term follow-up (week 6 months post-intervention)
  Ecologic Memory Simulations

SECONDARY OUTCOMES:
Changes in auditory processing speed | Baseline (week 1), immediately post-intervention (week 6) and long-term follow-up (week 6 months post-intervention)
  Paced Auditory Serial Edition Test
Changes in information processing speed | Baseline (week 1), immediately post-intervention (week 6) and long-term follow-up (week 6 months post-intervention)
  Symbol Digit Modalities Test
Changes in episodic verbal memory and learning | Baseline (week 1), immediately post-intervention (week 6) and long-term follow-up (week 6 months post-intervention)
  California Verbal Learning Test - 2nd Edition
Changes in visuospatial memory | Baseline (week 1), immediately post-intervention (week 6) and long-term follow-up (week 6 months post-intervention)
  Brief Visuospatial Memory Test - Revised
Changes in ability in spontaneous production of words | Baseline (week 1), immediately post-intervention (week 6) and long-term follow-up (week 6 months post-intervention)
  Controlled Oral Word Association Test
Changes in visual perception | Baseline (week 1), immediately post-intervention (week 6) and long-term follow-up (week 6 months post-intervention)
  Benton Judgment of Line Orientation
Changes in executive function | Baseline (week 1), immediately post-intervention (week 6) and long-term follow-up (week 6 months post-intervention)
  Delis-Kaplan Executive Function System - Sorting

CONTACTS AND LOCATIONS:
Overall Officials: Nancy D Chiaravalloti, PhD, Principal Investigator — Kessler Foundation
Locations (2):
- United States (2):
  - Kessler Foundation, East Hanover, New Jersey
  - Kessler Rehabilitation Center, Marlton, New Jersey

IPD SHARING:
Plan to Share IPD: No